CLINICAL TRIAL: NCT07134699
Title: The Impacts of Chronic Non-specific Low Back Pain on Cognitive Functions of Older Adults: A Longitudinal Study
Status: Recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, HSU Chun Liang, Assistant professor, The Hong Kong Polytechnic University
Other Study IDs: HSEARS20241003001
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-05

CONDITIONS: Chronic Non-Specific Low Back Pain; Cognitive Decline; Longitudinal Study; Older Adults; Brain Imaging
Keywords: Chronic Non-Specific low back pain; Cognitive decline; longitudinal study; older adults; brain imaging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic non-specific low back pain group: Participants with chronic non-specific low back pain (CNSLBP) should have: (1) CNSLBP that has lasted for at least 3 months, typically occurs in the area between the 12th rib to the iliac crest may or may not accompanied by leg pain and without a known pathoanatomical cause; (2) an average pain intensity of ≥ 5 out of 10 on an 11-point numerical rating scale (NRS) in the last 7 days, where 0 means "no pain"and 10 means "worst pain imaginable"; and (3) pain occurring more than 3 days per week.
  Interventions: Other: Participants are not assigned an intervention
- Healthy group: Healthy controls should not have CNSLBP in the last 36 months.
  Interventions: Other: Participants are not assigned an intervention

INTERVENTIONS:
Other: Participants are not assigned an intervention — For observational studies, participants are not assigned an intervention as part of the study.

SUMMARY:
Chronic non-specific low back pain (CNSLBP) is a common condition among older adults and has been associated with an increased risk of executive function impairment. Research shows that older adults experiencing chronic pain are more likely to show worse cognitive performance compared to healthy individuals. While there is a bidirectional relationship between pain and executive functions, cognitive performance especially for some executive functions (e.g. inhibition, switching, working memory) is crucial for managing pain in older adults. Furthermore, executive dysfunctions are associated with decline in functional status among the population, particularly in performing instrumental activities in daily living. Therefore, maintaining executive function emerges as a pivotal consideration for older adults with CNSLBP.

Studies provide preliminary evidence that connects brain changes with chronic pain and cognitive functions. For instance, multisite chronic pain may increase the risk of cognitive decline through structural changes like hippocampal atrophy. Besides, functional brain changes in chronic pain may reduce deactivation several key default mode network regions, predisposing individuals to cognitive impairments. Despite the aforementioned brain changes, no direct evidence supports the hypothesis that structural and functional brain changes caused by CNSLBP in older adults may be associated with cognitive decline. It remains unclear that whether structural changes (e.g. reduced hippocampal, cerebellar gray matter, white matter volume in the right frontal region) and/or functional changes (e.g. deactivation of default mode network regions, heightened activation in the anterior cingulate cortex) cause by CNSLBP are associated with cognitive decline. With neuroimaging techniques, brain mechanisms connecting CNSLBP and executive function deficits can be explained.

To deepen understanding of the brain mechanisms underlying executive function decline in older adults with CNSLBP, this study will directly compare pain intensity, executive functions, brain structure, and functional changes of the brain between older adults with CNSLBP and age-matched healthy controls. A longitudinal approach is established to quantify the relationship between CNSLBP-related brain changes and executive functions in older adults, providing insights into the development of new treatment strategies to improve or prevent executive function decline in older adults with CNSLBP.

ELIGIBILITY:
Inclusion Criteria:

* Older adults with and without chronic non-specific low back pain (CNSLBP) aged between 60 and 85 years
* Having normal cognitive function (Hong Kong Montreal Cognitive Assessment ≥ 26)13
* Right-handed
* Cantonese speaking
* Having at least 6 years of formal education and know how to read and write Chinese
* Agreeing to sign an informed consent form
* Being able to communicate via email or text message because several study measures will be collected electronically.

Exclusion Criteria:

* Inability to ambulate without assistance from another person (canes or walkers will be allowed)
* Having specific causes of LBP (e.g., spinal stenosis, lumbar disc herniation, spondylolisthesis, recent vertebral fracture, spinal infection)
* Having other concurrent musculoskeletal conditions at other body parts (e.g., fibromyalgia, or neck or knee pain)
* Self-reported history of lumbar or lower extremity surgery
* Self-reported history of neurological or psychiatric disorders (e.g., stroke, brain surgery, head trauma; schizophrenia, multiple personality disorder, dissociative identity disorder, stroke) or self-reported cancer history
* Self-reported specific inflammatory disorder: rheumatoid arthritis, rheumatica, scleroderma, lupus, or polymyositis
* Unexplained, unintended weight loss of 20 lbs or more in the past year
* Cauda equina syndrome
* Uncorrected visual deficit
* Drug or alcohol addiction
* Taking alcohol, opioids or benzodiazepines medicines 24 hours before the experiment
* Claustrophobia
* Contraindications for undergoing the magnetic resonance imaging (MRI) examination based on the MRI safety screening form of University Research Facility in Behavioral and Systems Neuroscience at The Hong Kong Polytechnic University

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with chronic non-specific low back pain (CNSLBP) should have:
  * CNSLBP that has lasted for at least 3 months, typically occurs in the area between the 12th rib to the iliac crest with and without leg pain and without a known pathoanatomical cause;
  * an average pain intensity of ≥ 5 out of 10 on an 11-point numerical rating scale (NRS) in the last 7 days, where 0 means "no pain" and 10 means "worst pain imaginable"; and
  * pain occurring more than 3 days per week. In addition, healthy controls should not have CNSLBP in the last 36 months.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity assessment | Baseline and 6 months
  11-point numerical rating scale, ranged from 0 to 10, higher scores indicate higher pain intensity.
Brain imaging | Baseline, 6 months
  Perform the following MRI sequences: T1-weighted, T2-weighted, DTI (diffusion tensor imaging), resting-state fMRI, and task-related fMRI.

SECONDARY OUTCOMES:
Depression, anxiety, and stress test | Baseline and 6 months
  The Chinese version of the short Depression Anxiety Stress Scales, scores ranged from 0 to 13, higher scores for each domain (depression, anxiety, and stress) indicate more respective problems.
Disability evaluation | Baseline and 6 months
  The Hong Kong Chinese Version of the Roland-Morris Disability Questionnaire has 24 items. Scores ranged from 0 to 24, higher scores indicate worse disability.
Cognitive flexibility test inside magnetic resonance imaging scanning | Baseline and 6 months
  The More Odd Shifting task, It requires participants to switch between different mental sets or rules, such as identifying odd numbers or shifting between different categories. Better response accuracy indicates better cognitive flexibility
Perseveration and abstract reasoning test outside magnetic resonance imaging scanning | Baseline and 6 months
  The Modified Wisconsin Card Sorting Test, more correct matching of cards indicate better perseveration and abstract reasoning.
Working memory Test outside magnetic resonance imaging scanning | Baseline and 6 months
  The Verbal Digits Forward and Backward Test, more correct recall of digits indicate better working memory and executive function
Cognitive flexibility test outside magnetic resonance imaging scanning | Baseline and 6 months
  The Trail Making Tests, a neuropsychological test of visual attention and task switching, completing the trail correctly within a shorter period of time means better cognitive flexibility.
Inhibition test outside magnetic resonance imaging scanning | Baseline and 6 months
  Go/NoGo task, more response accuracy indicates better control of inhibition.
Pain catastrophizing assessment | Baseline and 6 months
  The Chinese version of Pain Catastrophizing Score. The scores ranged from 0 to 13, higher scores indicate more pain catatrophizing thought.
Frailty status assessment | Baseline and 6 months
  Fatigue, Resistance, Ambulation, Illness, and Loss, the presence of 3 of 5 item characteristics indicate the presence of frailty, scores ranged from 0 to 5. Lower scores mean more frailty.
Sleep quality assessment | Baseline and 6 months
  Pittsburgh Sleep Quality Index. It has 7 domains to measure sleep quality , sleep latency, sleep duration, habital sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Scores ranged from 0 to 21, higher scores indicate poorer sleep quality.
Cognitive function screening | Baseline and 6 months
  Hong Kong Montreal Cognitive Assessment. It is a cognitive screening tool specifically adapted for Chinese older adults in Hong Kong. It is designed to detect mild cognitive impairment and dementia. A score < 26 suggests participant has mild cognitive impairment.
Balance, lower extremity strength and functional capacity assessment | Baseline and 6 months
  Short Physical Performance Battery (SPPB). It consists of three components: balance test, gait speed test, and chair stand test. The SPPB scores range from 0 to 12. Individuals with SPPB scores between 10 and 12 can exercise at home and in the community while those with more severe mobility limitations (scores < 10) require further assessment and supervision for exercise.
Mobility and balance assessment | Baseline and 6 months
  Timed Up and Go (TUG) test. It measures the time taken for an individual to rise from a chair, walk 3 meters, turn around, walk back, and sit down again. The TUG test helps identify individuals at risk of falls and mobility impairments. A shorter completion time indicates a better balance and functional mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Chun Liang Hsu, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Department of Rehabilitation Sciences, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided